CLINICAL TRIAL: NCT06396611
Title: Randomised Controlled Clinical Trial of Exercise As Intervention in Chronic Lymphocytic Leukemia
Brief Title: Exercise As Intervention in Chronic Lymphocytic Leukemia
Acronym: ADRENALINE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CLL_FADEUP
Record Dates: First submitted 2024-04-18; First posted 2024-05-02 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Strength Training; Physical Activity; Chronic Lymphocytic Leukemia; Vigorous Physical Activity
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Motor Activity | interventions — Exercise; Methods

STUDY DESIGN:
Intervention Model Description: Eligible patients who fulfil criteria will be randomized into a controlled design (RCT) comparing the effects of 16 weeks intervention program with a maximum of 2 sessions per week ensuring a 24h rest period between similar sessions, for the same aims and muscular groups. All participants are assessed in primary and secondary outcome measures before and after the intervention period. The intervention is designed with: a) Resistance Exercise Training (REX); b) Control Group (CG).
  We also expect to follow up those patients, after the intervention protocol terminus, using routine consultation on participating Hospitals, and acquiring data to support the long-term effects of the protocol. The follow-up will maintain the Onco-Hematology consultations routine and periodicity (6 months after last medical appointment), where all initial assessments will be undertaken.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Clinical evaluation is performed in invited hospitals, physical activity evaluation is performed by the outcomes assessor in Faculty of Sport of University of Porto. The investigator is the person who will conduct the intervention, and he's the one that will know what protocol is assigned to each patient, but without knowing the results from clinical and physical fitness evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistance Exercise Training (Experimental): Patients in the REx program are submitted to resistance machine exercises for the major muscle groups aiming to achieve the intensity of 80% of 1-Repetition Maximum (1-RM). A warmup and cool down of 10 and 5 minutes, respectively, were included in each session aiming workloads of 60%-85% of peak heart rate (HRp). Enrolment through the REx program resistance machines will be conducted from major muscle groups to minor muscle groups, from polyarticular to monoarticular exercises, and alternating between agonist and antagonist contraction according to the following laydown: Leg Press -> Leg Curl -> Leg Extension -> Chest Press -> Latissimus Pulldown -> Shoulder Press -> Triceps Extension -> Biceps Curl -> Abdominal Crunch.
  Interventions: Behavioral: Exercise Training as Intervention
- Conventional Care (Control Group) (No Intervention): Control group patients received advice to follow their habitual physical activity routines and are contacted bimonthly to ensure participant retention in the study.

INTERVENTIONS:
Behavioral: Exercise Training as Intervention — Supervised Exercise Training as an Intervention using Resistance Training.
  Arms: Resistance Exercise Training

SUMMARY:
PURPOSE: The purpose of the study is to determine the effects of 16-weeks of exercise training, as measured by aerobic capacity, strength and physical function, and body composition, in patients with Chronic Lymphocytic Leukemia (CLL).

DESIGN: Subjects will have confirmed treatment naïve CLL. Subjects will be assigned to either a 16-week control group (no supervised exercise) or an intervention group of Resistance Training (REx). Before and after the 16-week protocol, patients will undergo several tests including: 1) a maximal cycle ergometer test, 2) Body Composition, 3) Muscle strength, 4) physical activity levels, 5) blood measures (e.g. immune and inflammatory functions).

DATA ANALYSES & SAFETY ISSUES: For outcomes, group change differences from baseline to 16-weeks will be compared with ANCOVA. Resistance training is a very safe exercise modality already studied in other cancer patients. The regular use of vigorous-intensity exercise has been used extensively in exercise training. It will always be respected for each subject's safety tolerance while challenging.

HYPOTHESIS: The investigators hypothesize that the protocol will be feasible exercise interventions for people with CLL and will improve health and fitness markers.

DETAILED DESCRIPTION:
PURPOSE: The purpose of the study is to determine the effects of 16-weeks of exercise training, as measured by aerobic capacity, strength and physical function, and body composition, in patients with CLL and without any prior treatment.

DESIGN: Subjects will have confirmed treatment naïve CLL. Subjects will be assigned to either a 16-week control group (no supervised exercise) or an intervention group of Resistance Training (REx). Before and after the 16-week protocol, patients will undergo several tests including: 1) a Cardiopulmonary Exercise Test with Electrocardiogram (CPET+ECG) maximal cycle ergometer test, 2) a dual-energy X-ray absorptiometry (DEXA) Body Composition test, 3) a Muscle strength test with dynamometry, 4) a characterization of physical activity (PA) levels with accelerometry, and 5) blood measures (e.g. immune and inflammatory functions). The REx group will undertake a strength-based type of training with intensities near 80% of 1-Repetition Maximum (1-RM), with individual supervision (personal training approach).

DATA ANALYSES & SAFETY ISSUES: For outcomes, group change differences from baseline to 16-weeks will be compared with ANCOVA. Resistance training is a very safe exercise modality already studied in other cancer patients. The regular use of vigorous-intensity exercise has been used extensively in exercise training. It will always be respected for each subject's safety tolerance while challenging.

HYPOTHESIS: The investigators hypothesize that the protocol will be feasible exercise interventions for people with CLL and will improve health and fitness markers. It is also expected to have a positive correlation between physical fitness improvement and blood and immunologic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL as per the International Workshop on CLL Guidelines
* No history of previous treatment of CLL
* Able to walk on a treadmill or cycle ergometer
* Able to carry weights, or use weight machines
* Pass initial evaluations (CPET for cardiac health, Isokinetic for muscular health)
* Willing to adhere to the exercise program
* Signed informed consent

Exclusion Criteria:

* Previous CLL treatments
* Ongoing engagement in a regular exercise program
* Indication of disease progression and for starting treatment within 6 months
* Other primary tumour
* Inability to perform exercise (Heart disease, advanced stage respiratory, renal, hepatic, neurological, or osteoarticular disease)
* Unable to travel to FADEUP facilities or comply with other study requirements

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in VO2 peak as measured by cardiopulmonary exercise test | Baseline to 16-weeks
  Cardio metabolic CPET + Stress ECG
Change in muscular strength (peak torque and power) as measured by isokinetic dynamometer exercise test | Baseline to 16-weeks
  BIODEX Concentric/Concentric Strength Test for Lower Body evaluation
Change in muscular strength (grip force in kg) as measured by dynamometer exercise test | Baseline to 16-weeks
  JAMAR Hand Grip for Upper Body Evaluation
Change in muscular strength (kg of weight lifted) as measured by 1 repetition maximum exercise test | Baseline to 16-weeks
  1 Repetition Maximum For Strength Evaluation of Whole Body
Change in Whole Body Composition (comprehending grams of total mass, total fat mass, total lean mass and percentage of fat mass) | Baseline to 16-weeks
  DEXA Test for Whole Body Composition
Change in Bone Mineral Density (comprehending Total Femural and Femural Neck bone mineral density) | Baseline to 16-weeks
  DEXA Test for Bone Mineral Density

SECONDARY OUTCOMES:
Change in Health Related Quality of Life as measured by FACIT-F questionnaire | Baseline to 16-weeks
  Questionnaire The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F), a 40-item measure that assesses self-reported fatigue.
Change in Health Related Quality of Life as measured by EORTC QLQ-C30 and CLL17 questionnaires | Baseline to 16-weeks
  Questionnaire from EORTC Quality of Life Group (EORTC QLQ-C30) a 30-item instrument designed to measure quality of life in all cancer patients, with the supplement of CLL17 a 17-item instrument designed to measure quality of life in chronic lymphocytic leukemia patients
Change in Physical Activity patterns as measured by Accelerometry over a period of seven consecutive days | Baseline to 16-weeks
  GT9XLink accelerometer from Actigraph to collect data of the Physical Activity patterns, over a period of seven consecutive days, with a minimum of 10 hours of daily assessment
Change in Blood counts (hemoglobin (g/dL) and platelets (10^9/L)) as measured by Peripheral Blood Collection | Baseline to 16-weeks
  Peripheral Blood Collection during Hospital Consultation
Change in Leukocytes counts (in percentage of lymphocytes, monocytes, neutrophils) as measured by Peripheral Blood Collection | Baseline to 16-weeks
  Peripheral Blood Collection during Hospital Consultation
Change in Minerals counts (comprehending iron (ug/dL), sodium (mEq/L), potassium (mEq/L) and magnesium (mEq/L)) as measured by Peripheral Blood Collection | Baseline to 16-weeks
  Peripheral Blood Collection during Hospital Consultation

CONTACTS AND LOCATIONS:
Overall Officials: Pedro MP Cunha, MSc., Principal Investigator — Faculty of Sport of University of Porto
Locations (1):
- Faculty of Sport of University of Porto, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No
The datasets generated during the present study will not be publicly available, owing to the risk of disclosure or deduction of private individual information, but can be available from the corresponding author on reasonable request.